CLINICAL TRIAL: NCT05787743
Title: A Randomised Double-blinded Placebo Controlled Study on the Effect of Topical Palm Tocotrienol on Skin Biophysical Properties
Brief Title: Topical Palm Tocotrienols on Skin Biophysical Properties
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrawal
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Malaysia Palm Oil Board (Other Government); Avantsar Sdn. Bhd. (Unknown)
Responsible Party: Principal Investigator, Goh Choon Fu, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MA-T3-T1
Record Dates: First submitted 2023-02-17; First posted 2023-03-28 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Wrinkle
Keywords: tocotrienol; wrinkle; skin; topical; biophysical properties

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial cream with 2% palm tocotrienols extract (Active Comparator): Facial cream with 2% palm tocotrienols extract
  Interventions: Other: Facial cream with 2% palm tocotrienols extract
- Base cream (no active) (Placebo Comparator): Base cream (no active)
  Interventions: Other: Base cream

INTERVENTIONS:
Other: Facial cream with 2% palm tocotrienols extract — Apply on the face twice a day
  Arms: Facial cream with 2% palm tocotrienols extract
Other: Base cream — Apply on the face twice a day
  Arms: Base cream (no active)

SUMMARY:
A single-center, double-blind, randomised, placebo-controlled parallel-group study.

Selected subjects will be randomised into active and control groups in a ratio of 1:1. Investigational products assigned will be applied on the facial skin as part of daily skin care routine. The effects will be observed during the 24-weeks of use.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female individuals, aged 25 - 45 years old, inclusive
2. Fitzpatrick skin type II to IV
3. In generally good health and skin condition as determined by the PI or designee, based on medical history reported by the subject.
4. Willing to provide informed consent and comply with study procedures

Exclusion Criteria:

1. Has a history of chronic drug or alcohol abuse
2. Is current smoker
3. History of severe allergic reactions to topical products or vitamin E
4. Participant with severe and uncontrolled comorbidities (including but not limited to e.g. diabetes, hypertension, kidney failure)
5. Pregnant, breastfeeding, or planning pregnancy
6. Participant with known skin conditions (including but not limited to e.g. sensitive skin, eczema and diseased skin e.g. contact dermatitis), uncontrolled medical conditions, or any other condition that could interfere with the study evaluations or increase risk to the participant
7. Participant with compromised/broken skin, tattoos, scarring, excessive hair growth, very uneven skin tone, or other conditions that would interfere with evaluations or increase risk
8. Participation in another study within 4 weeks of screening visit

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 41 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in wrinkle (SEw) | 24 week
  Wrinkle

SECONDARY OUTCOMES:
Percent change from baseline in roughness (SEr), scaliness(SEsc), smoothness (SEsm), TEWL, Young's modulus, viscoelasticity, retraction time, collagen content, skin thickness, pigmentation index, erythema index, skin colour, pH, sebum and hydration | 24 week
  Skin biophysical properties
Percent change from baseline for Lemperle Wrinkle Assessment Scale | 24 week
  Wrinkle (scale 1 - 5; higher score for more wrinkles)
Percent change from baseline in scores of survey (BeautyQoL) | 24 week
  Survey (score 0 - 100%)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Pharmaceutical Sciences, Universiti Sains Malaysia, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi B, Heo JH, Kwon HJ, Lee ES, Sohn S. Tocotrienols enhance melanosome degradation through endosome docking/fusion proteins in B16F10 melanoma cells. Food Funct. 2013 Oct;4(10):1481-8. doi: 10.1039/c3fo60289c. PMID 23995710
- [Background] Chu CC, Hasan ZABA, Tan CP, Nyam KL. In Vitro Antiaging Evaluation of Sunscreen Formulated from Nanostructured Lipid Carrier and Tocotrienol-Rich Fraction. J Pharm Sci. 2021 Dec;110(12):3929-3936. doi: 10.1016/j.xphs.2021.08.020. Epub 2021 Aug 21. PMID 34425132
- [Background] Draize, J.H., Woodard, G., Calvery, H.O., 1944. Methods for the study of irritation and toxicity of substances applied topically to the skin and mucous membranes. Journal of Pharmacology and Experimental Therapeutics 82, 377-390.
- [Background] Harun MS, Wong TW, Fong CW. Advancing skin delivery of alpha-tocopherol and gamma-tocotrienol for dermatitis treatment via nanotechnology and microwave technology. Int J Pharm. 2021 Jan 25;593:120099. doi: 10.1016/j.ijpharm.2020.120099. Epub 2020 Nov 28. PMID 33259902
- [Background] Ikeda S, Niwa T, Yamashita K. Selective uptake of dietary tocotrienols into rat skin. J Nutr Sci Vitaminol (Tokyo). 2000 Jun;46(3):141-3. doi: 10.3177/jnsv.46.141. PMID 10955281
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Makpol S, Abidin AZ, Sairin K, Mazlan M, Top GM, Ngah WZ. gamma-Tocotrienol prevents oxidative stress-induced telomere shortening in human fibroblasts derived from different aged individuals. Oxid Med Cell Longev. 2010 Jan-Feb;3(1):35-43. doi: 10.4161/oxim.3.1.9940. PMID 20716926
- [Background] Mei Yee, C., Ahmad, N., Azizul Hasan, Z.A., Abu Hasan, H., 2014. Tocotrienol-Based Facial Masks, MPOB Information Series. Malaysian Palm Oil Board, Kuala Lumpur, Malaysia.
- [Background] Muggli R. Systemic evening primrose oil improves the biophysical skin parameters of healthy adults. Int J Cosmet Sci. 2005 Aug;27(4):243-9. doi: 10.1111/j.1467-2494.2005.00274.x. PMID 18492193
- [Background] Musalmah M, Nizrana MY, Fairuz AH, NoorAini AH, Azian AL, Gapor MT, Wan Ngah WZ. Comparative effects of palm vitamin E and alpha-tocopherol on healing and wound tissue antioxidant enzyme levels in diabetic rats. Lipids. 2005 Jun;40(6):575-80. doi: 10.1007/s11745-005-1418-9. PMID 16149736
- [Background] Patel V, Rink C, Gordillo GM, Khanna S, Gnyawali U, Roy S, Shneker B, Ganesh K, Phillips G, More JL, Sarkar A, Kirkpatrick R, Elkhammas EA, Klatte E, Miller M, Firstenberg MS, Chiocca EA, Nesaretnam K, Sen CK. Oral tocotrienols are transported to human tissues and delay the progression of the model for end-stage liver disease score in patients. J Nutr. 2012 Mar;142(3):513-9. doi: 10.3945/jn.111.151902. Epub 2012 Feb 1. PMID 22298568
- [Background] Pedrelli VF, Lauriola MM, Pigatto PD. Clinical evaluation of photoprotective effect by a topical antioxidants combination (tocopherols and tocotrienols). J Eur Acad Dermatol Venereol. 2012 Nov;26(11):1449-53. doi: 10.1111/j.1468-3083.2011.04219.x. Epub 2011 Sep 14. PMID 21917024
- [Background] Sen CK, Khanna S, Roy S. Tocotrienols in health and disease: the other half of the natural vitamin E family. Mol Aspects Med. 2007 Oct-Dec;28(5-6):692-728. doi: 10.1016/j.mam.2007.03.001. Epub 2007 Mar 27. PMID 17507086
- [Background] Shibata A, Nakagawa K, Kawakami Y, Tsuzuki T, Miyazawa T. Suppression of gamma-tocotrienol on UVB induced inflammation in HaCaT keratinocytes and HR-1 hairless mice via inflammatory mediators multiple signaling. J Agric Food Chem. 2010 Jun 9;58(11):7013-20. doi: 10.1021/jf100691g. PMID 20465215
- [Background] Suzuki YJ, Tsuchiya M, Wassall SR, Choo YM, Govil G, Kagan VE, Packer L. Structural and dynamic membrane properties of alpha-tocopherol and alpha-tocotrienol: implication to the molecular mechanism of their antioxidant potency. Biochemistry. 1993 Oct 12;32(40):10692-9. doi: 10.1021/bi00091a020. PMID 8399214
- [Background] Thiele JJ, Traber MG, Podda M, Tsang K, Cross CE, Packer L. Ozone depletes tocopherols and tocotrienols topically applied to murine skin. FEBS Lett. 1997 Jan 20;401(2-3):167-70. doi: 10.1016/s0014-5793(96)01463-9. PMID 9013880
- [Background] Thiele JJ, Traber MG, Tsang K, Cross CE, Packer L. In vivo exposure to ozone depletes vitamins C and E and induces lipid peroxidation in epidermal layers of murine skin. Free Radic Biol Med. 1997;23(3):385-91. doi: 10.1016/s0891-5849(96)00617-x. PMID 9214574
- [Background] Traber MG, Podda M, Weber C, Thiele J, Rallis M, Packer L. Diet-derived and topically applied tocotrienols accumulate in skin and protect the tissue against ultraviolet light-induced oxidative stress. Asia Pac J Clin Nutr. 1997 Mar;6(1):63-7. PMID 24394657
- [Background] Tsuduki T, Kuriyama K, Nakagawa K, Miyazawa T. Tocotrienol (unsaturated vitamin E) suppresses degranulation of mast cells and reduces allergic dermatitis in mice. J Oleo Sci. 2013;62(10):825-34. doi: 10.5650/jos.62.825. PMID 24088520
- [Background] Yamada Y, Obayashi M, Ishikawa T, Kiso Y, Ono Y, Yamashita K. Dietary tocotrienol reduces UVB-induced skin damage and sesamin enhances tocotrienol effects in hairless mice. J Nutr Sci Vitaminol (Tokyo). 2008 Apr;54(2):117-23. doi: 10.3177/jnsv.54.117. PMID 18490840
- [Background] Yamashita, E., 2006. Cosmetic benefit of dietary supplements including astaxanthin and tocotrienol on human skin.
- [Background] Yap WN. Tocotrienol-rich fraction attenuates UV-induced inflammaging: A bench to bedside study. J Cosmet Dermatol. 2018 Jun;17(3):555-565. doi: 10.1111/jocd.12421. Epub 2017 Sep 26. PMID 28952200
- [Background] Yap WN, Zaiden N, Xu CH, Chen A, Ong S, Teo V, Yap YL. Gamma- and delta-tocotrienols inhibit skin melanin synthesis by suppressing constitutive and UV-induced tyrosinase activation. Pigment Cell Melanoma Res. 2010 Oct;23(5):688-92. doi: 10.1111/j.1755-148X.2010.00740.x. Epub 2010 Jul 27. No abstract available. PMID 20609176
- [Background] Yusuf, N.Z., Azizul Hasan, Z.A., Ismail, R., 2011. TOCOGELS As Anti-Inflammatory Agents, MPOB Information Series. Malaysian Palm Oil Board, Kuala Lumpur, Malaysia.
- [Background] Zainal Z, Khaza'ai H, Kutty Radhakrishnan A, Chang SK. Therapeutic potential of palm oil vitamin E-derived tocotrienols in inflammation and chronic diseases: Evidence from preclinical and clinical studies. Food Res Int. 2022 Jun;156:111175. doi: 10.1016/j.foodres.2022.111175. Epub 2022 Mar 21. PMID 35651097